CLINICAL TRIAL: NCT06278766
Title: Mass Balance Study of [14C] ABBV-552 in Healthy Male Volunteers Following Single Oral Dose Administration
Brief Title: A Study to Assess the Mass Balance of [14C] ABBV-552 in Healthy Male Participants Following Single Oral Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M24-416
Record Dates: First submitted 2024-02-20; First posted 2024-02-26 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-552

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-552 (Experimental): Participants will receive ABBV-552 on Day 1.
  Interventions: Drug: ABBV-552

INTERVENTIONS:
Drug: ABBV-552 — Oral Solution

SUMMARY:
The purpose of this study is to evaluate mass balance, pharmacokinetics and safety of [14C] ABBV-552 in healthy, male volunteers following administration of a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

- Male volunteers in general good health at Screening.

Exclusion Criteria:

- Considering fathering a child or donating sperm during the study and for 100 days after study drug administration.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 30 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum observed concentration (Cmax) of ABBV-552 | Up to approximately Day 15
  Cmax of ABBV-552 will be assessed.
Time to Cmax (peak time, Tmax) of ABBV-552 | Up to approximately 15 days
  Tmax of ABBV-552 will be assessed.
Terminal phase elimination rate constant (λz) of ABBV-552 | Up to approximately 15 days
  Terminal phase elimination rate constant (λz) of ABBV-552 will be assessed.
Terminal phase elimination half-life (t1/2) of ABBV-552 | Up to approximately 15 days
  Terminal phase elimination half-life (t1/2) of ABBV-552 will be assessed.
Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration (AUCt) of ABBV-552 | Up to approximately 15 days
  AUCt of ABBV-552 will be assessed.
Area under the plasma concentration-time curve (AUC) from time 0 to infinite time (AUCinf) of ABBV-552 | Up to approximately 15 days
  AUCinf of ABBV-552 will be assessed.
Amount of ABBV-552 excreted in the urine over the sampling period (Aeu) | Up to approximately 15 days
  Amount of ABBV-552 excreted in the urine over the sampling period (Aeu) will be assessed.
Percent of ABBV-552 excreted in the urine | Up to approximately 15 days
  Percent excreted = 100 × (Aeu/dose).
Renal clearance ABBV-552 (CLr) | Up to approximately 15 days
  Renal clearance of ABBV-552 will be assessed.
Amount of ABBV-552 excreted in the feces over the sampling period (Aef) | Up to approximately 15 days
  Amount of ABBV-552 excreted in the feces over the sampling period (Aef) will be assessed.
Percent radioactivity excreted in the feces | Up to approximately 15 days
  Percent excreted = 100 × (Aef/dose).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Fortrea Clinical Research Unit Inc /ID# 262684, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-416